CLINICAL TRIAL: NCT01348750
Title: Healing Touch and Guided Imagery Intervention in Post-deployment Military Personnel With Posttraumatic Stress Disorder Symptoms
Brief Title: Healing Touch & Guided Imagery for Posttraumatic Stress Disorder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Center for Integrative Medicine (Other)
Collaborators: Marine Corps Base Camp Pendleton (Other)
Responsible Party: Erminia M. Guarneri, MD, Medical Director, Scripps Center for Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTSD_HSC07_4684
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Healing Touch; Guided Imagery; Military; Complementary Medicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Touch; Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): This group receives 6 Healing Touch & Guided Imagery treatments in addition to standard medical care.
  Interventions: Other: Healing Touch & Guided Imagery
- Group B (No Intervention): This group receives standard medical care but NO Healing Touch and Guided Imagery.

INTERVENTIONS:
Other: Healing Touch & Guided Imagery — Healing Touch (HT) is an energy based approach to health and healing. It uses light touch to influence the energy field that surrounds the body, and the energy centers which control the flow of energy to the physical body.
  HT complements traditional health care and is used together with other approaches to health and healing.
  Guided Imagery (GI) is a form of focused relaxation used to create harmony between the mind and body. Positive mental imagery can promote relaxation, reduce stress and improve mood as well as alter heart rate, blood pressure and breathing.
  Arms: Group A

SUMMARY:
This is a randomized controlled 2 year trial at Camp Pendleton, CA to determine whether a complementary medicine intervention (Healing Touch with Guided Imagery, HT+GI) reduces Posttraumatic Stress Disorder (PTSD) symptoms as compared to treatment as usual (TAU) in returning combat-exposed active duty military with significant PTSD symptoms. Secondary aims will evaluate the effect of HT and GI on measures of depression, hostility, and general health status in this population.

DETAILED DESCRIPTION:
The study enrolled 123 active duty subjects from the Marine Corps Base Camp Pendleton in Southern California with at least one or more symptoms of PTSD .

ELIGIBILITY:
Inclusion Criteria:

1. Female or male subjects 18 years or older
2. Post-deployment from a combat zone
3. Identified by post-deployment health re-assessment to have PTSD symptoms
4. Referred by Camp Pendleton
5. Subjects who are willing to sign a consent
6. Subjects who are willing to participate for the length of the study

Exclusions:

1. Female subjects who are now pregnant or nursing
2. Subjects who are receiving healing touch or using guided imagery from other sources
3. Subjects who have any major health condition that may interfere with participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
17-item PTSD Checklist (Military)is used to determine the effect of the intervention | After 6 treatments of healing touch and guided imagery

SECONDARY OUTCOMES:
Depression (Beck Depression Inventory) | After 6 treatments of healing touch and guided imagery
Quality of Life (SF36) | After 6 treatments of healing touch and guided imagery
Hostility (Cook-Medley Hostility Inventory) | After 6 treatments of healing touch and guided

CONTACTS AND LOCATIONS:
Overall Officials: Erminia M Guarneri, MD, Principal Investigator — Scripps Center for Integrative Medicine
Locations (1):
- Scripps Center for Integrative Medicine, La Jolla, California, United States